CLINICAL TRIAL: NCT01159886
Title: Patient-posture and Ileal-intubation During Colonoscopy (PIC): a Randomized Controlled Open-label Trial
Brief Title: Patient-posture and Ileal-intubation During Colonoscopy
Acronym: PIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Dr Kshaunish Das, Associate Professor, Division of Gastroenterology, SDLD, IPGME & R, Kolkata-700020
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SDLD001
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Colonoscopy
Keywords: Tuberculosis; IBD; endoscopy
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- left lateral (Active Comparator): After confirmation of cecal intubation, patient will undergo randomization to either the left-lateral decubitus position. Then terminal ileal intubation will be attempted.
  Interventions: Procedure: Ileal intubation
- supine (Active Comparator): After confirmation of cecal intubation, patient will undergo randomization to the supine position. Then terminal ileal intubation will be attempted.
  Interventions: Procedure: Ileal intubation

INTERVENTIONS:
Procedure: Ileal intubation — After confirmation of cecal intubation, patient will undergo randomization to either the left-lateral decubitus or supine position. Then terminal ileal intubation will be attempted. Partial suction and scope manoeuvres for ileal intubation will be allowed.
  Use of anti-peristalsis agents, use of biopsy forceps, as a guidewire or an ''anchor'' to facilitate the IC- valve intubation, and intubation in the retroflexed position will not be allowed.
  Other Names: Ileoscopy

SUMMARY:
During colonoscopy, the colonoscopist employs various maneuvers, including changing the patient's posture to left-lateral decubitus or supine, to achieve complete colonoscopic examination. Posture change has also been reported to increase the success rate of ileal intubation. However, there has been no randomized trial which has shown that a particular posture of the patient increases the success rate of ileoscopy. The present study will be carried out to determine the impact of the patient's posture (left lateral vs supine position) on success rate of ileal intubation.

ELIGIBILITY:
Inclusion Criteria:

* All adult (> 12y old) patients referred for colonoscopy

Exclusion Criteria:

* Acute fulminant colitis
* Acute Intestinal obstruction
* Suspected intestinal perforation
* Peritonitis
* Pregnancy
* Severe cardio-respiratory disease (ASA grade…)
* Decompensated liver disease
* Recent pelvic or colonic surgery (in last 6 months)
* Large aortic or ileac artery aneurysm
* Human Immunodeficiency Virus Infection
* Uncooperative patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-01 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Ileal intubation achieved or not | After confirmation of cecal intubation for no more than 6 minutes
  After confirmation of cecal intubation, patient will undergo randomization to either the left-lateral decubitus or supine position. Then terminal ileal intubation will be attempted. Two points will be assessed: success in ileal intubation and time taken to intubate the ileum. If ileum is not intubated within 6 minutes, it will be considered as failed attempt.

SECONDARY OUTCOMES:
Time taken to intubate the ileum after cecal intubation | 6 minutes after cecal intubation and randomisation
Depth of ileal intubation | 2 minutes
Influence of endoscopist experience on successful ileal intubation | 6 minutes
Abnormal ileal findings | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kshaunish Das, MD, DM, Principal Investigator — Associate Professor, Division of Gastroenterology, SDLD, IPGME & R, Kolkata-700020
Locations (1):
- School of Digestive and Liver Diseases (SDLD), IPGME & R, Kolkata, Kolkata, India